CLINICAL TRIAL: NCT00582478
Title: Investigating Mechanisms to Explain Age Associated Differences in Quality of Life Among Breast Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Wake Forest University (Other)
Responsible Party: Sponsor
Other Study IDs: 01-120
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Reproductive History; Weights and Measures; prostacyclin synthetase; Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: women with breast cancer
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Participants will be followed regularly at 3, 6, 12, and 18-month intervals
  Other Names: Functional Assessment of Cancer Therapy - Fact B, 2. Beck Depression Inventory, 3. MOS Sexual Functioning; Questionnaire, 4. Body Appearance Scale, 5. SF-36 Health Status Questionnaire, 6.; Global Quality of Life, 7. Interval Medical and Reproductive History, 8. Physical; Symptoms Checklist, 9. RAND Social Support Scale, 10. Funtional Assessment of; Chronic Illness Therapy-Spiritual Well Being (FACIT-Sp) 11.Optimisim, 12 Brief COPE; Scale, 13. Illness Intrusive Scale, 14. Posttraumatic Growth Inventory (PTGI), 15.; Quality of Life in Adult Cancer Survivors (QLACS).

SUMMARY:
The purpose of this study is to look at how breast cancer treatment affects quality of life in women of different ages. The U.S. Army Breast Cancer Research Program funds this study. In this research project, we wish to study a woman's quality of life after breast cancer treatment as related to her health. We want to know how you feel about your quality of life.

DETAILED DESCRIPTION:
This multi-center study will include self-referred. This project is a prospective cohort study of 800 women aged 18 and over who are newly diagnosed with breast cancer. Women will be recruited into the study within 6 months after diagnosis and followed for 18 months. The primary purpose of the proposed study is to examine mechanisms that may explain age differences in the health-related quality of life of women who have been diagnosed with a first-time breast cancer. The studies will examine psychosocial factors such as social support, coping strategies, resiliency, and the impact of cancer on life responsibilities as explanations of age-associated factors affecting HRQL. This project is an observational, longitudinal study of women aged 18 and over who are newly diagnosed with breast cancer. In order to examine both the short- and longer-term impact of breast cancer on HRQL, the study will survey women post diagnosis and follow them at 3, 6, 12, and 18 months. A secondary purpose is to have this large cohort of breast cancer patients serve as a comparison group for other studies in the Behavioral Center of Excellence award given to Wake Forest Medical Center by the Department of Defense. Extensive baseline data will be collected by an in-depth chart review and interview for additional data. Information will be gathered on demographics, clinical and treatment variables. The study intervention consists of collecting data on health-related quality of life through specific questionnaires.

Data collection instruments will be mailed to participants at regularly scheduled intervals accompanied by a stamped,addressed envelope. If the participant does not return study forms within three weeks, the participant will be called.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 or older at the time of breast cancer diagnosis
* English-speaking
* Community dwelling (i.e. not living in a residential care or correctional facility)
* Diagnosed with invasive breast cancer Stage I, II, or III within the previous 6 months
* First time diagnosis
* Have physician agreement for participation
* Provide informed consent

Exclusion Criteria:

* Psychiatric or psychological abnormality precluding informed consent or ability to complete questionnaires
* Previous or concurrent malignancy (except basal and squamous skin cancer and stage 0 cervical cancer)
* Stage IV breast malignancy
* Residency outside of the United States
* For women ages 45 years and younger only: Those participants < 45 years who were having regular menstrual cycles at the time of diagnosis will be excluded from this protocol. This study will only be enrolling women in this age category who have had a prior hysterectomy or were having irregular menstrual cycles at the time of diagnosis. Women with regular menstrual cycles will be enrolled into a companion project (i.e., Menstrual Cycle Maintenance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First time breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2001-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The study measurements are quality of life questionnaires | 7 years 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Tracy-Ann Moo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org